CLINICAL TRIAL: NCT02032446
Title: UMBILICAL CORD DERIVED MESENCHYMAL STROMAL CELLS (UC-MSC) FOR THE TREATMENT OF SEVERE (GRADE III-IV) STEROID-RESISTANT GRAFT VERSUS HOST DISEASE (GvHD): A PHASE I/II TRIAL
Brief Title: Umbilical Cord Derived Mesenchymal Stromal Cells For The Treatment of Severe Steroid-resistant Graft Versus Host Disease
Acronym: PTC-UC-MSC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Principal Investigator, Rambaldi Alessandro, Head Hematology and Bone Marrow Transplant Unit, A.O. Ospedale Papa Giovanni XXIII
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2012-000582-21
Record Dates: First submitted 2013-11-04; First posted 2014-01-10 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical Cord Mesenchymal stromal cells (UC-MSC) (Experimental): Pentostatin will be given by intravenous infusion at a dose of 1 mg/m2 for 3 consecutive days. Thereafter, three Umbilical Cord Mesenchymal stromal cells (UC-MSC) infusions will be given at weekly interval starting from day 5. We will follow a dose escalating programme with progressively increasing doses of cells until the maximally tolerated dose (MTD) is achieved.
  The dose escalating design will be characterised by the administration of 1x106 /kg UC-MSC per dose per three doses for the first three patients (total up to 3x106/kg). The second three patients will receive 2x106/kg UC-MSC per dose per three doses (total up to 6x106/kg). The third three patients will receive 3x106/kg UC-MSC per dose per three doses (total up to 9x106 cells/kg).
  Since three dosages of cells are programmed for each group of 3 patients, a minimum of 9 patients should be studied, unless unacceptable acute infusion related toxicity is observed.
  Interventions: Biological: UMBILICAL CORD DERIVED MESENCHYMAL STROMAL CELLS (UC-MSC)

INTERVENTIONS:
Biological: UMBILICAL CORD DERIVED MESENCHYMAL STROMAL CELLS (UC-MSC) — pentostatin, dose 1 mg/m2
  § MSC doses:
  1. 3 patients → 3 infusions of 1x106 cells /kg
  2. 3 patients → 3 infusions of 2x106 cells /kg
  3. 3 patients → 3 infusions of 3x106 cells /kg

SUMMARY:
MESENCHYMAL STROMAL CELLS (MSC) have shown promising albeit not always consistent therapeutic effects in the treatment of severe steroid-resistant acute Graf versus Host Disease. Remarkably, in all reported clinical studies the toxicity of Mesenchymal stromal cells administration has been found consistently negligible. The investigators believe that Umbilical Cord (UC) derived Mesenchymal stromal cells may represent a stronger immunosuppressive tool for such clinical emergency and no data suggest any change in the safety profile of these cells. For this reason, and in the best interest of the patient, the investigators plan to test the safety and activity of Umbilical Cord Mesenchymal stromal cells when given sequentially to another partially effective treatment of steroid resistant acute graf versus host disease such as Pentostatin.

ELIGIBILITY:
Inclusion Criteria:

Patients are required to meet the following inclusion criteria:

1. Patients with steroid refractory grade III-IV classic acute graft versus host disease (GvHD)occurring within 100 days after transplant or induced by donor lymphocyte infusions (DLI) or T-cell add back. Steroid refractory graft versus host disease (GvHD)is defined according to Pidala and Anasetti10 as follows: a) progression of at least 1 overall grade within 3 days of optimal steroid treatment; b) failure to demonstrate any overall grade improvement over 5 to 7 days; c) incomplete response by 14 days of 2 mg/kg/day of steroid therapy.
2. Patients with persistent, recurrent, or late acute graft versus host disease (GvHD) (features of acute graft versus host disease occurring beyond 100 days, often during withdrawal of immune suppression).
3. Patients with an overlap syndrome in which diagnostic or distinctive features of chronic graft versus host disease (GvHD) and acute graft versus host disease (GvHD) appear together79.

Exclusion Criteria:

1. Inability to obtain written informed consent

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
vital parameters | one year
  Following infusion of UC-MSC, the patient will be monitored for acute infusion-related toxicity. Any toxicity will be treated at the discretion of the attending physician. Infusional toxicity is defined as any alteration of the vital parameters of the patient if they have appeared acutely and may be directly correlated to the UC-MSC infusion

SECONDARY OUTCOMES:
assessed of acute graft versus host disease (GvHD) | one year
  graft versus host disease will be assessed at day +7, +9, +12, +14, +16, +19, +21, +28, + 35, +42 e +49 and after 6 months and 1 year from the last UC-MSC infusion. Efficacy on acute graft versus host disease is defined as complete or partial resolution of acute GvHD evaluated according to conventional staging and grading score systems.The efficacy will be evaluated at day +30 after the third UC-MSC infusion or, if less, at day +30 after the last UC-MSC infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rambaldi, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII
Locations (8):
- Italy (8):
  - A O Papa Giovanni XXIII, Bergamo
  - Ao S Croce E Carle, Cuneo
  - AO Careggi, Florence
  - IRCCS G Gaslini, Genova
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Clinica Pediatrica San Gerardo, Monza
  - Azienda Ospedaliero-Universitaria Di Udine, Udine
  - Ospedale San Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: Yes
interim analysis

REFERENCES:
- [Result] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Result] Capelli C, Gotti E, Morigi M, Rota C, Weng L, Dazzi F, Spinelli O, Cazzaniga G, Trezzi R, Gianatti A, Rambaldi A, Golay J, Introna M. Minimally manipulated whole human umbilical cord is a rich source of clinical-grade human mesenchymal stromal cells expanded in human platelet lysate. Cytotherapy. 2011 Aug;13(7):786-801. doi: 10.3109/14653249.2011.563294. Epub 2011 Mar 18. PMID 21417678
- [Result] Lucchini G, Introna M, Dander E, Rovelli A, Balduzzi A, Bonanomi S, Salvade A, Capelli C, Belotti D, Gaipa G, Perseghin P, Vinci P, Lanino E, Chiusolo P, Orofino MG, Marktel S, Golay J, Rambaldi A, Biondi A, D'Amico G, Biagi E. Platelet-lysate-expanded mesenchymal stromal cells as a salvage therapy for severe resistant graft-versus-host disease in a pediatric population. Biol Blood Marrow Transplant. 2010 Sep;16(9):1293-301. doi: 10.1016/j.bbmt.2010.03.017. Epub 2010 Mar 27. PMID 20350611
- [Result] Ringden O, Uzunel M, Rasmusson I, Remberger M, Sundberg B, Lonnies H, Marschall HU, Dlugosz A, Szakos A, Hassan Z, Omazic B, Aschan J, Barkholt L, Le Blanc K. Mesenchymal stem cells for treatment of therapy-resistant graft-versus-host disease. Transplantation. 2006 May 27;81(10):1390-7. doi: 10.1097/01.tp.0000214462.63943.14. PMID 16732175
- [Result] von Bonin M, Stolzel F, Goedecke A, Richter K, Wuschek N, Holig K, Platzbecker U, Illmer T, Schaich M, Schetelig J, Kiani A, Ordemann R, Ehninger G, Schmitz M, Bornhauser M. Treatment of refractory acute GVHD with third-party MSC expanded in platelet lysate-containing medium. Bone Marrow Transplant. 2009 Feb;43(3):245-51. doi: 10.1038/bmt.2008.316. Epub 2008 Sep 29. PMID 18820709
- [Result] Perez-Simon JA, Lopez-Villar O, Andreu EJ, Rifon J, Muntion S, Diez Campelo M, Sanchez-Guijo FM, Martinez C, Valcarcel D, Canizo CD. Mesenchymal stem cells expanded in vitro with human serum for the treatment of acute and chronic graft-versus-host disease: results of a phase I/II clinical trial. Haematologica. 2011 Jul;96(7):1072-6. doi: 10.3324/haematol.2010.038356. Epub 2011 Mar 10. PMID 21393326
- [Result] Weiss ML, Anderson C, Medicetty S, Seshareddy KB, Weiss RJ, VanderWerff I, Troyer D, McIntosh KR. Immune properties of human umbilical cord Wharton's jelly-derived cells. Stem Cells. 2008 Nov;26(11):2865-74. doi: 10.1634/stemcells.2007-1028. Epub 2008 Aug 14. PMID 18703664
- See also: Agenzia Italiana del Farmaco (AIFA) — http://www.agenziafarmaco.gov.it